CLINICAL TRIAL: NCT01923233
Title: Phase I Feasibility Study of ALLOSTIM(TM) in Combination With Radiofrequency Ablation in Patients With Refractory Hepatocellular Carcinoma
Brief Title: In-Situ Therapeutic Cancer Vaccine for Refractory Liver Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: interventional radiologist suffered stroke and unable to perform RFA procedure
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-017-HCC
Record Dates: First submitted 2013-08-12; First posted 2013-08-15 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2015-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; HCC; tumor vaccine; immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Intradermal AlloStim(TM) (1ml) on day 0 and 3 in same location Intradermal AlloStim(TM) (1ml) on day 7 and day 10 in same location Radiofrequency ablation on day 14 followed by intralesional AlloStim (3ml) Intralesional AlloStim(TM)(3ml) on day 17 in same ablated lesion Intravenous AlloStim(TM)(5ml) on days 21, 49 and 78
  Interventions: Biological: AlloStim

INTERVENTIONS:
Biological: AlloStim — allogeneic Th1 memory cell with CD3/CD28-coated microbeads attached.
  Other Names: InSituVax

SUMMARY:
This study is an individualized anti-cancer vaccine protocol where the vaccination occurs inside of the body. To create the vaccine, a tumor lesion is selected and caused to die by a process called "Radiofrequency Ablation" or RFA. RFA causes the tumor to release its internal contents to the surrounding environment, such contents include tumor-specific antigens. Immune cells respond to the tissue damage and take-up these tumor antigens. The injection of the experimental cell drug, AlloStim(TM) into the lesion is designed to cause the responding cells to signal the immune system of the danger of the tumor, creating tumor-specific immunity.

DETAILED DESCRIPTION:
The protocol design has 4 steps: (1) priming; (2) vaccination, (3) activation and (4) boosting. The priming step involves intradermal injections of AlloStim(TM). This is designed to increase the circulating titer of allo-specific Th1 memory cells; the vaccination step involves percutaneous radiofrequency ablation of a single liver lesion followed immediately with an intratumoral injection of AlloStim(TM) into the ablated lesion, followed 3 days later by an additional intratumoral injection into the previously ablated lesion with AlloStim(TM). This step is designed to elicit tumor-specific Th1 immunity. The activation step involves intravenous infusions of AlloStim(TM). This step is designed to cause the activation and extravasation of circulating memory cells and the activation of innate immune cells. The booster step includes two monthly IV infusions of AlloStim(TM). This step is designed to maintain an inflammatory cytokine storm designed to counteract immune suppressor mechanisms and tumor immunoavoidance mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Any patients with a diagnosis of HCC based on histology or the current accepted radiological measures.
2. Age > 18 years.
3. Patient has an MRI or CT result (positive for HCC) up to 3 months prior to recruitment.
4. AFP >30.
5. Patient who is not eligible for or failed any HCC treatment.

Exclusion Criteria:

1. Patient is unable or unwilling to sign informed consent.
2. Patients that are participating in other clinical trials evaluating experimental treatments or procedures
3. Severe congestive heart failure (LVEF on echocardiogram < 20%).
4. Severe pulmonary hypertension (By echocardiogram, PAS >45 mmHg).
5. Uncontrolled diabetes mellitus (HBA1C >9.5%).
6. Any autoimmune disorder, which is currently being treated with prednisone or any other immune suppressive medication.
7. Patients currently receiving total parenteral nutrition if they have contraindications to oral drugs.
8. Subjects with positive HIV.
9. Women who are pregnant or breast feeding.
10. Patient, based on the opinion of the investigator, should not be enrolled into this study.
11. HBsAg positive or HBV DNA positive.
12. If the patient is HBcAB positive but HBsAG negative, irrespective of his anti HBS status, he can be enrolled but will receive preemptive therapy with Lamivudine.
13. Any metastasis except for portal vein involvement.
14. Subjects with Child Pugh above B8.
15. Prior experimental therapy or cancer vaccine treatment (e.g., dendritic cell therapy, heat shock vaccine).
16. History of blood transfusion reactions.
17. Known allergy to bovine or murine products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Safety | baseline to 90 days
  Subjects will be followed by physical exam, blood labs, CT scan and biopsy for any adverse events

SECONDARY OUTCOMES:
Tumor-Specific Immunity | 90 days
  Determine if the in-situ vaccine elicits detectable tumor specific immunity
Anti-Tumor Response | 90 days
  Determine by radiological, pathological, immunological and by tumor markers any evidence of anti-tumor immune-mediated response.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Har-Noy, Study Director — Mirror Biologics, Inc.
Locations (1):
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Epple LM, Bemis LT, Cavanaugh RP, Skope A, Mayer-Sonnenfeld T, Frank C, Olver CS, Lencioni AM, Dusto NL, Tal A, Har-Noy M, Lillehei KO, Katsanis E, Graner MW. Prolonged remission of advanced bronchoalveolar adenocarcinoma in a dog treated with autologous, tumour-derived chaperone-rich cell lysate (CRCL) vaccine. Int J Hyperthermia. 2013 Aug;29(5):390-8. doi: 10.3109/02656736.2013.800997. Epub 2013 Jun 20. PMID 23786302
- [Background] Mayer-Sonnenfeld T, Har-Noy M, Lillehei KO, Graner MW. Proteomic analyses of different human tumour-derived chaperone-rich cell lysate (CRCL) anti-cancer vaccines reveal antigen content and strong similarities amongst the vaccines along with a basis for CRCL's unique structure: CRCL vaccine proteome leads to unique structure. Int J Hyperthermia. 2013 Sep;29(6):520-7. doi: 10.3109/02656736.2013.796529. Epub 2013 Jun 4. PMID 23734882
- [Background] LaCasse CJ, Janikashvili N, Larmonier CB, Alizadeh D, Hanke N, Kartchner J, Situ E, Centuori S, Har-Noy M, Bonnotte B, Katsanis E, Larmonier N. Th-1 lymphocytes induce dendritic cell tumor killing activity by an IFN-gamma-dependent mechanism. J Immunol. 2011 Dec 15;187(12):6310-7. doi: 10.4049/jimmunol.1101812. Epub 2011 Nov 9. PMID 22075702
- [Background] Janikashvili N, LaCasse CJ, Larmonier C, Trad M, Herrell A, Bustamante S, Bonnotte B, Har-Noy M, Larmonier N, Katsanis E. Allogeneic effector/memory Th-1 cells impair FoxP3+ regulatory T lymphocytes and synergize with chaperone-rich cell lysate vaccine to treat leukemia. Blood. 2011 Feb 3;117(5):1555-64. doi: 10.1182/blood-2010-06-288621. Epub 2010 Dec 1. PMID 21123824
- [Background] Har-Noy M, Zeira M, Weiss L, Fingerut E, Or R, Slavin S. Allogeneic CD3/CD28 cross-linked Th1 memory cells provide potent adjuvant effects for active immunotherapy of leukemia/lymphoma. Leuk Res. 2009 Apr;33(4):525-38. doi: 10.1016/j.leukres.2008.08.017. Epub 2008 Oct 1. PMID 18834631
- [Background] Har-Noy M, Slavin S. The anti-tumor effect of allogeneic bone marrow/stem cell transplant without graft vs. host disease toxicity and without a matched donor requirement? Med Hypotheses. 2008;70(6):1186-92. doi: 10.1016/j.mehy.2007.10.008. Epub 2007 Dec 3. PMID 18054441